CLINICAL TRIAL: NCT03422159
Title: Outcomes of Metabolic Resuscitation Using Ascorbic Acid, Thiamine, and Glucocorticoids in the Early Treatment of Sepsis.
Brief Title: Metabolic Resuscitation Using Ascorbic Acid, Thiamine, and Glucocorticoids in Sepsis.
Acronym: ORANGES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Community Medical Center, Toms River, NJ (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17-004
Record Dates: First submitted 2018-01-25; First posted 2018-02-05 (Actual); Results first posted 2021-09-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2020-11

CONDITIONS: Sepsis, Severe; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Ascorbic Acid; Thiamine; Hydrocortisone; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This is a double-blind placebo controlled study. Only the dispensing pharmacist will be aware of the treatment allocation. Patients will be randomized to receive either vitamin C/hydrocortisone/thiamine or triple placebo using a random number table provided to the dispensing pharmacists. Each patient will be allocated a unique subject ID which will be linked to the randomization sequence. Only the dispensing pharmacists will have a record of the subject ID and randomization sequence.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients will be randomized to receive either vitamin C/hydrocortisone/thiamine or triple placebo using a random number table provided to the dispensing pharmacists. Each patient will be allocated a unique subject ID which will be linked to the randomization sequence. Only the dispensing pharmacists will have a record of the subject ID and randomization sequence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Experimental): Based on published clinical data, vitamin C pharmacokinetic modeling, the package insert as well as the preliminary study by Marik et al, Vitamin C will be administered as an intravenous dose of 6gm per day divided in 4 equal doses. This dosage is reported to be devoid of any complications or side effects. Hydrocortisone will be dosed according to the consensus guidelines of the American College of Critical Care Medicine. Thiamine will be administered according to current recommendations in a dose of 200mg q 12 hourly. This will be continued for 4 days, or less if discharged from the ICU prior.
  Interventions: Drug: Ascorbic Acid; Drug: Thiamine; Drug: Hydrocortisone
- Placebo Arm (Placebo Comparator): Vitamin C placebo will consist of an identical bag of 100mL normal saline (but with no vitamin C) and will be labeled "Vitamin C or Placebo". Placebo will be infused over 30 minutes as per the infusion instructions of the active vitamin and protected from light with a brown bag. Hydrocortisone placebo will be provided as an identical 3mL syringe as 1mL of normal saline.The thiamine placebo will be placed in a 50mL bag of Normal Saline labeled "Thiamine 200mg or Placebo" and run over 30 minutes (100mL/hr) Placebo patients will receive a matching 50mL bag of Normal Saline. All of these will be given for up to 4 days, or less if discharged from the ICU prior.
  Interventions: Drug: Sodium Chloride 0.9%

INTERVENTIONS:
Drug: Ascorbic Acid — Ascorbic Acid 1.5g IV piggyback every 6 hours for 4 days (or discharge from ICU if prior to 4 days).
  Other Names: Vitamin C
  Arms: Treatment Arm
Drug: Thiamine — Thiamine 200mg IV piggyback every 12 hours for 4 days (or discharge from ICU if prior to 4 days).
  Arms: Treatment Arm
Drug: Hydrocortisone — Hydrocortisone 50mg IV push every 6 hours for 4 days (or discharge from ICU if prior to 4 days).
  Other Names: Solucortef
  Arms: Treatment Arm
Drug: Sodium Chloride 0.9% — Placebo "Ascorbic Acid" 100mL IV piggyback every 6 hours, Placebo "Thiamine" 50mL IV piggyback every 12 hours, and Placebo "Hydrocortisone" IV push every 6 hours for 4 days (or discharge from ICU if prior to 4 days).
  Other Names: Placebo
  Arms: Placebo Arm

SUMMARY:
This study has been created to compare the addition of intravenous (IV) vitamin C, thiamine, and hydrocortisone to the usual standard of care of sepsis and septic shock. Sepsis is a possibly life-threatening condition in which a patient may have organ dysfunction due to an infection. Septic shock is defined as low blood pressure and organ dysfunction that do not improve after administering IV fluids. Standard of care for sepsis and septic shock include early administration of IV antibiotics, IV fluids, and vasopressors if need be to provide oxygen to vital organs.

A large amount of experimental data has shown that vitamin C and corticosteroids decrease the release of inflammatory substances which may lead to organ failure seen in sepsis. Vitamin C and corticosteroids also improve blood flow to vital organs and increase the body's ability to respond well to vasopressor medications used in septic shock. Low blood levels of both thiamine and vitamin C are common in sepsis. The study will be placebo controlled, meaning one group will receive vitamin C, thiamine, and hydrocortisone, and the other will receive an inactive substance ("placebo"). The goal of the study is to compare the effects of receiving vitamin C, thiamine, and hydrocortisone (along with the standard sepsis care) versus placebo and standard sepsis care.

DETAILED DESCRIPTION:
The global burden of sepsis is substantial with an estimated 15 to 19 million cases per year; the vast majority of these cases occur in low income countries. With more timely diagnosis and improvement in supportive care the 28-day mortality from sepsis in high income countries has declined to about 25%, however, the mortality from septic shock remains as high as 45%. Moreover, the mortality from sepsis and septic shock in low income countries is reported to be as high as 60%. In addition to short term mortality, septic patients suffer from a numerous short- and long-term complications and are at an increased risk of death for up to five years following the acute event. Over the last 3 decades over 100 phase II and phase III clinical trial have been performed testing various novel pharmacologic agents and therapeutic intervention in an attempt to improve the outcome of patients with sepsis and septic shock; all of these studies have failed to show an improvement in patient outcomes. New therapeutic approaches to sepsis are desperately required; considering the global burden of sepsis these interventions should be effective, cheap, safe and readily available.

A large body of experimental data has demonstrated that both corticosteroids and intravenous vitamin C reduce activation of nuclear factor ƘB (NFƘB) attenuating the release of pro-inflammatory mediators, reduce the endothelial injury characteristic of sepsis thereby reducing endothelial permeability and improving macrocirculatory flow, augment the release of endogenous catecholamines and enhance vasopressor responsiveness. In animal models these effects have resulted in reduced organ injury and increased survival. Corticosteroids have been evaluated in several clinical trials, with meta-analysis of these trials demonstrating somewhat conflicting outcomes. Low-dose stress corticosteroids have proven to be safe with no increased risk of clinically important complications. While corticosteroids decrease vasopressor dependency the effect on survival is less clear.

Several studies have investigated the use of intravenous vitamin C in critically ill patients. Nathens et al randomized 595 surgical ICU patients (91% trauma patients) to receive intravenous vitamin C and vitamin E for up to 28 days.The vitamin combination was associated with a significant reduction in the incidence of multiple system organ failure (p=0.04) with a trend to reduced mortality and length of ICU stay. No adverse effects were noted with the vitamin combination. Fowler et al performed a pilot study in 24 patients with severe sepsis and septic shock. In this study patients were randomized to placebo (n=8), low dose intravenous vitamin C (50 mg/kg) (n=8) or high dose vitamin C (200mg/kg). Vitamin C attenuated the inflammatory response with both doses of the vitamin being devoid of any side effects. Although the Sequential Sepsis Related Organ Failure Score (SOFA) fell significantly in both treatment arms the study was underpowered to determine any outcome benefit. Zabet and colleagues performed a randomized controlled trial (RCT) in which they evaluated the role of intravenous vitamin C in a dose of 100 mg/kg/day (about 7g/day) in 28 surgical ICU patients with septic shock. In this study the mean dose of norepinephrine and duration of norepinephrine administration were significantly lower in the ascorbic acid than the placebo group. The 28-day mortality was significantly lower in the ascorbic acid than the placebo group (14% vs. 64%, p = 0.009). No side effects related to the vitamin C infusion were reported. Tanaka et al randomized 37 patients with severe burn to very high dose vitamin C (about 110g/day) or placebo. Patients who received vitamin C required less fluid resuscitation with a trend towards reduced length of stay and mortality. No adverse effects were noted with the very high dosages of vitamin C. Several studies have administered vitamin C in doses exceeding 100g/day as adjuvant therapy in patients with cancer with no discernable side effects. Vitamin C appears to be toxic to normal human cells (not cancer cells) at a concentration on greater than 25 millimole (mM). A dose of 6g/day will achieve a steady state serum concentration of about 240 micromole (uM) which is about 100 times less than the dose required to cause cellular toxicity. The package insert for vitamin C lists no contraindications or adverse effects of the drug and states that as much as "6 grams has been administered without evidence of toxicity". The only reported restriction to the use of high dose intravenous vitamin C is in patients with known glucose-6-phosphate deficiency (G6PD) in whom hemolysis has been reported. It is important to recognize that patents with sepsis predictably have very low serum vitamin C levels, which can only be corrected with intravenous vitamin C in a dose of more than 3gm per day. The low or undetectable levels of vitamin C likely result from the metabolic consumption of the molecule as well as increased renal losses. Furthermore, unlike all other mammals, primates and guinea pigs are unable synthesize vitamin C is due to mutations in the L-gulono-_-lactone oxidase (GLO) gene which codes for the enzyme responsible for catalyzing the last step of vitamin C biosynthesis. In almost all species, except humans and guinea pigs, vitamin C production increases during stress and is secreted by the adrenal gland; in these species vitamin C is best considered a stress "hormone". Vitamin C is an essential cofactor for the production of corticosteroids and catecholamines by the adrenal gland. Vitamin C has been shown to reverse adrenal suppression caused by induction doses of etomidate during anesthesia.

Ascorbate donates a single electron in all its redox reactions, generating the ascorbate radical. This radical is not very reactive with anything but itself. Dismutation of two ascorbate radicals forms a molecule each of ascorbate and dehydroascorbate. Hydrolysis of the lactone ring of dehydroascorbate irreversibly converts it to 2,3-diketo-1-gulonic acid which is then converted to oxalate. Oxalate is normally excreted by the kidney and serum levels will increase with renal impairment. In patients with renal impairment receiving mega-dose vitamin C, supersaturation of serum with oxalate may result in tissue deposition as well as crystallization in the kidney. Glyoxylate, a byproduct of intermediary metabolism, is either reduced to oxalate or oxidized to carbon dioxide (CO2) by the enzyme glyoxylate aminotransferase; thiamine pyrophosphate is a co-enzyme required for this reaction. Thiamine deficiency increases the conversion of glyoxylate to oxalate resulting in hyper- oxalosis. Donnino and colleagues have demonstrated that thiamine deficiency is common (32%) in patients with sepsis and that treatment with thiamine in these patients reduces mortality. In a post-hoc analysis of this study these authors demonstrated that thiamine decreased the risk of acute kidney injury and the required for renal replacement therapy in all treated patients.

It has previously been suggested that "...the best hope for therapeutic advances [in sepsis] will depend on broad-base targeting, in which multiple components are targeted at the same time." Such combination "chemo-therapy" targeting multiple biological pathways is the standard approach in the treatment of malignant disease. While the benefits of vitamin C, hydrocortisone, and thiamine alone are likely limited, the investigators believe that these medications act synergistically to reduce the risk of organ failure and death in patients with sepsis. This hypothesis is supported previous research and more recently a set of elegant experiments performed by Barabutis et al. Using a validated pulmonary endothelial monolayer model, these authors demonstrated that hydrocortisone together with vitamin C protected the vascular endothelium from damage by endotoxin while neither agent alone had this effect. Previous research has demonstrated that vitamin C reverses oxidation of the glucocorticoid receptor (GR) a likely manifestation of sepsis. Oxidation of the GR limits binding of the GR to both ligand and DNA responsive units decreasing the activity of glucocorticoids. Furthermore, glucocorticoids increase the expression of the sodium vitamin C transporter-2 (SVCT-2) which is an essential transport protein necessary for vitamin C to be transported intracellularly.

The investigators therefore propose that a "metabolic resuscitation protocol" including vitamin C, corticosteroids and thiamine will limit the development of organ failure and reduce mortality in patients with severe sepsis and septic shock. This postulate is supported by the preliminary findings by Marik et al. In a retrospective before-after clinical study, these authors compared the outcome and clinical course of consecutive septic patients treated with intravenous vitamin C, hydrocortisone and thiamine during a 7-month period (treatment group) compared to a control group treated in during the preceding 7 months. The primary outcome was hospital survival. A propensity score was generated to adjust the primary outcome. There were 47 patients in both treatment and control groups with no significant differences in baseline characteristics between the two groups. The hospital mortality was 8.5% (4 of 47) in the treatment group compared to 40.4% (19 of 47) in the control group (p < 0.001). The propensity adjusted odds of mortality in the patients treated with the vitamin C protocol was 0.13 (95% CI 0.04-0.48, p=0.002). The SOFA score decreased in all patients in the treatment group with none developing progressive organ failure. Vasopressors were weaned off all patients in the treatment group, a mean of 18.3 ± 9.8 hours after starting treatment with vitamin C protocol. The mean duration of vasopressor use was 54.9 ± 28.4 hours in the control group (p<0.001). The results of this study provide sufficient information for the design of an adequately powered, pragmatic randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

i. Diagnosis of sepsis or septic shock within 12 hours of admission to the ICU ii. Informed consent as dictated by IRB and local practice. iii. Compliance with the 3 hour sepsis bundle

* 30ml/kg of intravenous crystalloid fluid (e.g.: sodium chloride 0.9%) for lactic acid >4 and/or systolic blood pressure <90mmHg / mean arterial pressure <65mmHg
* Lactic acid level drawn
* Broad spectrum antibiotics given after obtaining blood cultures

Exclusion Criteria:

i. Age < 18 years ii. Pregnant iii. DNR/DNI with limitations of care on admission iv. Patients with terminal end stage disease (i.e. stage IV cancer, end stage heart failure) that are unlikely to survive to hospital discharge v. Patients with a primary admitting diagnosis of an acute cerebral vascular event, acute coronary syndrome, active gastrointestinal bleeding, burn or trauma [64-66] vi. Requirement for immediate surgery [64-66] vii. Patients with HIV and a CD4 < 50 mm2 [64-66] viii. Patients with known glucose-6 phosphate dehydrogenase (G-6PD) deficiency.[39] ix. Patients with sepsis/septic shock transferred from another hospital x. Patients with features of sepsis/septic shock > 24 hours after admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-08-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Monmouth Medical Center, Southern Campus, Lakewood, New Jersey
  - Community Medical Center, Toms River, New Jersey

REFERENCES:
- [Background] Adhikari NK, Fowler RA, Bhagwanjee S, Rubenfeld GD. Critical care and the global burden of critical illness in adults. Lancet. 2010 Oct 16;376(9749):1339-46. doi: 10.1016/S0140-6736(10)60446-1. Epub 2010 Oct 11. PMID 20934212
- [Background] Kaukonen KM, Bailey M, Suzuki S, Pilcher D, Bellomo R. Mortality related to severe sepsis and septic shock among critically ill patients in Australia and New Zealand, 2000-2012. JAMA. 2014 Apr 2;311(13):1308-16. doi: 10.1001/jama.2014.2637. PMID 24638143
- [Background] Silva E, Pedro Mde A, Sogayar AC, Mohovic T, Silva CL, Janiszewski M, Cal RG, de Sousa EF, Abe TP, de Andrade J, de Matos JD, Rezende E, Assuncao M, Avezum A, Rocha PC, de Matos GF, Bento AM, Correa AD, Vieira PC, Knobel E; Brazilian Sepsis Epidemiological Study. Brazilian Sepsis Epidemiological Study (BASES study). Crit Care. 2004 Aug;8(4):R251-60. doi: 10.1186/cc2892. Epub 2004 Jun 15. PMID 15312226
- [Background] Sales Junior JA, David CM, Hatum R, Souza PC, Japiassu A, Pinheiro CT, Friedman G, Silva OB, Dias MD, Koterba E, Dias FS, Piras C, Luiz RR; Grupo de Estudo de Sepse do Fundo AMIB. [An epidemiological study of sepsis in Intensive Care Units: Sepsis Brazil study]. Rev Bras Ter Intensiva. 2006 Mar;18(1):9-17. Portuguese. PMID 25310321
- [Background] The 10 leading causes of death by country income group 2012. WHO factsheets. http://www.who.int/mediacentre/factsheets/fs310/en/index1.html . 2015. World Health Organization. 5-24-2016.
- [Background] Wang HE, Szychowski JM, Griffin R, Safford MM, Shapiro NI, Howard G. Long-term mortality after community-acquired sepsis: a longitudinal population-based cohort study. BMJ Open. 2014 Jan 17;4(1):e004283. doi: 10.1136/bmjopen-2013-004283. PMID 24441058
- [Background] Artenstein AW, Higgins TL, Opal SM. Sepsis and scientific revolutions. Crit Care Med. 2013 Dec;41(12):2770-2. doi: 10.1097/CCM.0b013e31829eb98f. PMID 23989175
- [Background] Fisher BJ, Seropian IM, Kraskauskas D, Thakkar JN, Voelkel NF, Fowler AA 3rd, Natarajan R. Ascorbic acid attenuates lipopolysaccharide-induced acute lung injury. Crit Care Med. 2011 Jun;39(6):1454-60. doi: 10.1097/CCM.0b013e3182120cb8. PMID 21358394
- [Background] Fisher BJ, Kraskauskas D, Martin EJ, Farkas D, Puri P, Massey HD, Idowu MO, Brophy DF, Voelkel NF, Fowler AA 3rd, Natarajan R. Attenuation of sepsis-induced organ injury in mice by vitamin C. JPEN J Parenter Enteral Nutr. 2014 Sep;38(7):825-39. doi: 10.1177/0148607113497760. Epub 2013 Aug 5. PMID 23917525
- [Background] Han M, Pendem S, Teh SL, Sukumaran DK, Wu F, Wilson JX. Ascorbate protects endothelial barrier function during septic insult: Role of protein phosphatase type 2A. Free Radic Biol Med. 2010 Jan 1;48(1):128-35. doi: 10.1016/j.freeradbiomed.2009.10.034. Epub 2009 Oct 17. PMID 19840845
- [Background] Kim SR, Ha YM, Kim YM, Park EJ, Kim JW, Park SW, Kim HJ, Chung HT, Chang KC. Ascorbic acid reduces HMGB1 secretion in lipopolysaccharide-activated RAW 264.7 cells and improves survival rate in septic mice by activation of Nrf2/HO-1 signals. Biochem Pharmacol. 2015 Jun 15;95(4):279-89. doi: 10.1016/j.bcp.2015.04.007. Epub 2015 Apr 17. PMID 25896849
- [Background] Bornstein SR, Yoshida-Hiroi M, Sotiriou S, Levine M, Hartwig HG, Nussbaum RL, Eisenhofer G. Impaired adrenal catecholamine system function in mice with deficiency of the ascorbic acid transporter (SVCT2). FASEB J. 2003 Oct;17(13):1928-30. doi: 10.1096/fj.02-1167fje. Epub 2003 Aug 1. PMID 12897061
- [Background] Wilson JX. Mechanism of action of vitamin C in sepsis: ascorbate modulates redox signaling in endothelium. Biofactors. 2009 Jan-Feb;35(1):5-13. doi: 10.1002/biof.7. PMID 19319840
- [Background] Wilson JX. Evaluation of vitamin C for adjuvant sepsis therapy. Antioxid Redox Signal. 2013 Dec 10;19(17):2129-40. doi: 10.1089/ars.2013.5401. Epub 2013 Jun 25. PMID 23682970
- [Background] Marik PE. Critical illness-related corticosteroid insufficiency. Chest. 2009 Jan;135(1):181-193. doi: 10.1378/chest.08-1149. PMID 19136406
- [Background] Annane D, Bellissant E, Bollaert PE, Briegel J, Keh D, Kupfer Y. Corticosteroids for treating sepsis. Cochrane Database Syst Rev. 2015 Dec 3;2015(12):CD002243. doi: 10.1002/14651858.CD002243.pub3. PMID 26633262
- [Background] Minneci PC, Deans KJ, Eichacker PQ, Natanson C. The effects of steroids during sepsis depend on dose and severity of illness: an updated meta-analysis. Clin Microbiol Infect. 2009 Apr;15(4):308-18. doi: 10.1111/j.1469-0691.2009.02752.x. PMID 19416302
- [Background] Kalil AC, Sun J. Low-dose steroids for septic shock and severe sepsis: the use of Bayesian statistics to resolve clinical trial controversies. Intensive Care Med. 2011 Mar;37(3):420-9. doi: 10.1007/s00134-010-2121-0. Epub 2011 Jan 18. PMID 21243334
- [Background] Sprung CL, Annane D, Keh D, Moreno R, Singer M, Freivogel K, Weiss YG, Benbenishty J, Kalenka A, Forst H, Laterre PF, Reinhart K, Cuthbertson BH, Payen D, Briegel J; CORTICUS Study Group. Hydrocortisone therapy for patients with septic shock. N Engl J Med. 2008 Jan 10;358(2):111-24. doi: 10.1056/NEJMoa071366. PMID 18184957
- [Background] Nathens AB, Neff MJ, Jurkovich GJ, Klotz P, Farver K, Ruzinski JT, Radella F, Garcia I, Maier RV. Randomized, prospective trial of antioxidant supplementation in critically ill surgical patients. Ann Surg. 2002 Dec;236(6):814-22. doi: 10.1097/00000658-200212000-00014. PMID 12454520
- [Background] Fowler AA 3rd, Syed AA, Knowlson S, Sculthorpe R, Farthing D, DeWilde C, Farthing CA, Larus TL, Martin E, Brophy DF, Gupta S; Medical Respiratory Intensive Care Unit Nursing; Fisher BJ, Natarajan R. Phase I safety trial of intravenous ascorbic acid in patients with severe sepsis. J Transl Med. 2014 Jan 31;12:32. doi: 10.1186/1479-5876-12-32. PMID 24484547
- [Background] Zabet MH, Mohammadi M, Ramezani M, Khalili H. Effect of high-dose Ascorbic acid on vasopressor's requirement in septic shock. J Res Pharm Pract. 2016 Apr-Jun;5(2):94-100. doi: 10.4103/2279-042X.179569. PMID 27162802
- [Background] Tanaka H, Matsuda T, Miyagantani Y, Yukioka T, Matsuda H, Shimazaki S. Reduction of resuscitation fluid volumes in severely burned patients using ascorbic acid administration: a randomized, prospective study. Arch Surg. 2000 Mar;135(3):326-31. doi: 10.1001/archsurg.135.3.326. PMID 10722036
- [Background] Ma Y, Chapman J, Levine M, Polireddy K, Drisko J, Chen Q. High-dose parenteral ascorbate enhanced chemosensitivity of ovarian cancer and reduced toxicity of chemotherapy. Sci Transl Med. 2014 Feb 5;6(222):222ra18. doi: 10.1126/scitranslmed.3007154. PMID 24500406
- [Background] Hoffer LJ, Robitaille L, Zakarian R, Melnychuk D, Kavan P, Agulnik J, Cohen V, Small D, Miller WH Jr. High-dose intravenous vitamin C combined with cytotoxic chemotherapy in patients with advanced cancer: a phase I-II clinical trial. PLoS One. 2015 Apr 7;10(4):e0120228. doi: 10.1371/journal.pone.0120228. eCollection 2015. PMID 25848948
- [Background] Hoffer LJ, Levine M, Assouline S, Melnychuk D, Padayatty SJ, Rosadiuk K, Rousseau C, Robitaille L, Miller WH Jr. Phase I clinical trial of i.v. ascorbic acid in advanced malignancy. Ann Oncol. 2008 Nov;19(11):1969-74. doi: 10.1093/annonc/mdn377. Epub 2008 Jun 9. PMID 18544557
- [Background] Stephenson CM, Levin RD, Spector T, Lis CG. Phase I clinical trial to evaluate the safety, tolerability, and pharmacokinetics of high-dose intravenous ascorbic acid in patients with advanced cancer. Cancer Chemother Pharmacol. 2013 Jul;72(1):139-46. doi: 10.1007/s00280-013-2179-9. Epub 2013 May 14. PMID 23670640
- [Background] Monti DA, Mitchell E, Bazzan AJ, Littman S, Zabrecky G, Yeo CJ, Pillai MV, Newberg AB, Deshmukh S, Levine M. Phase I evaluation of intravenous ascorbic acid in combination with gemcitabine and erlotinib in patients with metastatic pancreatic cancer. PLoS One. 2012;7(1):e29794. doi: 10.1371/journal.pone.0029794. Epub 2012 Jan 17. PMID 22272248
- [Background] Welsh JL, Wagner BA, van't Erve TJ, Zehr PS, Berg DJ, Halfdanarson TR, Yee NS, Bodeker KL, Du J, Roberts LJ 2nd, Drisko J, Levine M, Buettner GR, Cullen JJ. Pharmacological ascorbate with gemcitabine for the control of metastatic and node-positive pancreatic cancer (PACMAN): results from a phase I clinical trial. Cancer Chemother Pharmacol. 2013 Mar;71(3):765-75. doi: 10.1007/s00280-013-2070-8. Epub 2013 Feb 5. PMID 23381814
- [Background] Ohno S, Ohno Y, Suzuki N, Soma G, Inoue M. High-dose vitamin C (ascorbic acid) therapy in the treatment of patients with advanced cancer. Anticancer Res. 2009 Mar;29(3):809-15. PMID 19414313
- [Background] de Grooth HJ, Choo WP, Spoelstra-de Man AM et al. Pharmacokinetics of four high- dose regimens of intravenous Vitamin C in critically ill patients [Abstract]. Intensive Care Med 2016.
- [Background] Padayatty SJ, Sun H, Wang Y, Riordan HD, Hewitt SM, Katz A, Wesley RA, Levine M. Vitamin C pharmacokinetics: implications for oral and intravenous use. Ann Intern Med. 2004 Apr 6;140(7):533-7. doi: 10.7326/0003-4819-140-7-200404060-00010. PMID 15068981
- [Background] Long CL, Maull KI, Krishnan RS, Laws HL, Geiger JW, Borghesi L, Franks W, Lawson TC, Sauberlich HE. Ascorbic acid dynamics in the seriously ill and injured. J Surg Res. 2003 Feb;109(2):144-8. doi: 10.1016/s0022-4804(02)00083-5. PMID 12643856
- [Background] Ascorbic Acid Injection. http://www.drugs.com/pro/ascorbic-acid-injection.html . 2015. The Torrance Company. 6-12-2016.
- [Background] Campbell GD Jr, Steinberg MH, Bower JD. Letter: Ascorbic acid-induced hemolysis in G-6-PD deficiency. Ann Intern Med. 1975 Jun;82(6):810. doi: 10.7326/0003-4819-82-6-810_1. No abstract available. PMID 1138591
- [Background] Rees DC, Kelsey H, Richards JD. Acute haemolysis induced by high dose ascorbic acid in glucose-6-phosphate dehydrogenase deficiency. BMJ. 1993 Mar 27;306(6881):841-2. doi: 10.1136/bmj.306.6881.841. No abstract available. PMID 8490379
- [Background] Drouin G, Godin JR, Page B. The genetics of vitamin C loss in vertebrates. Curr Genomics. 2011 Aug;12(5):371-8. doi: 10.2174/138920211796429736. PMID 22294879
- [Background] Patak P, Willenberg HS, Bornstein SR. Vitamin C is an important cofactor for both adrenal cortex and adrenal medulla. Endocr Res. 2004 Nov;30(4):871-5. doi: 10.1081/erc-200044126. PMID 15666839
- [Background] Das D, Sen C, Goswami A. Effect of Vitamin C on adrenal suppression by etomidate induction in patients undergoing cardiac surgery: A randomized controlled trial. Ann Card Anaesth. 2016 Jul-Sep;19(3):410-7. doi: 10.4103/0971-9784.185522. PMID 27397444
- [Background] Nooraei N, Fathi M, Edalat L et al. Effect of Vitamin C on serum cortisol after etomidate induction of anesthesia. J Cell Mol Anesth 2016; 1:28-33.
- [Background] Massey LK, Liebman M, Kynast-Gales SA. Ascorbate increases human oxaluria and kidney stone risk. J Nutr. 2005 Jul;135(7):1673-7. doi: 10.1093/jn/135.7.1673. PMID 15987848
- [Background] Wandzilak TR, D'Andre SD, Davis PA, Williams HE. Effect of high dose vitamin C on urinary oxalate levels. J Urol. 1994 Apr;151(4):834-7. doi: 10.1016/s0022-5347(17)35100-5. PMID 8126804
- [Background] Hoppe B, Beck BB, Milliner DS. The primary hyperoxalurias. Kidney Int. 2009 Jun;75(12):1264-1271. doi: 10.1038/ki.2009.32. Epub 2009 Feb 18. PMID 19225556
- [Background] Sidhu H, Gupta R, Thind SK, Nath R. Oxalate metabolism in thiamine-deficient rats. Ann Nutr Metab. 1987;31(6):354-61. doi: 10.1159/000177294. PMID 3426152
- [Background] Ortiz-Alvarado O, Miyaoka R, Kriedberg C, Moeding A, Stessman M, Monga M. Pyridoxine and dietary counseling for the management of idiopathic hyperoxaluria in stone-forming patients. Urology. 2011 May;77(5):1054-8. doi: 10.1016/j.urology.2010.08.002. Epub 2011 Feb 19. PMID 21334732
- [Background] Donnino MW, Andersen LW, Chase M, Berg KM, Tidswell M, Giberson T, Wolfe R, Moskowitz A, Smithline H, Ngo L, Cocchi MN; Center for Resuscitation Science Research Group. Randomized, Double-Blind, Placebo-Controlled Trial of Thiamine as a Metabolic Resuscitator in Septic Shock: A Pilot Study. Crit Care Med. 2016 Feb;44(2):360-7. doi: 10.1097/CCM.0000000000001572. PMID 26771781
- [Background] Moskowitz A, Andersen LW, Cocchi MN, Karlsson M, Patel PV, Donnino MW. Thiamine as a Renal Protective Agent in Septic Shock. A Secondary Analysis of a Randomized, Double-Blind, Placebo-controlled Trial. Ann Am Thorac Soc. 2017 May;14(5):737-741. doi: 10.1513/AnnalsATS.201608-656BC. PMID 28207287
- [Background] Aird WC. The role of the endothelium in severe sepsis and multiple organ dysfunction syndrome. Blood. 2003 May 15;101(10):3765-77. doi: 10.1182/blood-2002-06-1887. Epub 2003 Jan 23. PMID 12543869
- [Background] Marik PE, Pastores SM, Annane D, Meduri GU, Sprung CL, Arlt W, Keh D, Briegel J, Beishuizen A, Dimopoulou I, Tsagarakis S, Singer M, Chrousos GP, Zaloga G, Bokhari F, Vogeser M; American College of Critical Care Medicine. Recommendations for the diagnosis and management of corticosteroid insufficiency in critically ill adult patients: consensus statements from an international task force by the American College of Critical Care Medicine. Crit Care Med. 2008 Jun;36(6):1937-49. doi: 10.1097/CCM.0b013e31817603ba. PMID 18496365
- [Background] Okamoto K, Tanaka H, Makino Y, Makino I. Restoration of the glucocorticoid receptor function by the phosphodiester compound of vitamins C and E, EPC-K1 (L-ascorbic acid 2-[3,4-dihydro-2,5,7,8-tetramethyl-2-(4,8,12-trimethyltridecyl)-2H-1-benzopyran-6-yl hydrogen phosphate] potassium salt), via a redox-dependent mechanism. Biochem Pharmacol. 1998 Jul 1;56(1):79-86. doi: 10.1016/s0006-2952(98)00121-x. PMID 9698091
- [Background] Fujita I, Hirano J, Itoh N, Nakanishi T, Tanaka K. Dexamethasone induces sodium-dependant vitamin C transporter in a mouse osteoblastic cell line MC3T3-E1. Br J Nutr. 2001 Aug;86(2):145-9. doi: 10.1079/bjn2001406. PMID 11502226
- [Background] Barabutis N, Khangoora V, Marik PE, Catravas JD. Hydrocortisone and Ascorbic Acid Synergistically Prevent and Repair Lipopolysaccharide-Induced Pulmonary Endothelial Barrier Dysfunction. Chest. 2017 Nov;152(5):954-962. doi: 10.1016/j.chest.2017.07.014. Epub 2017 Jul 21. PMID 28739448
- [Background] Marik PE, Khangoora V, Rivera R, Hooper MH, Catravas J. Hydrocortisone, Vitamin C, and Thiamine for the Treatment of Severe Sepsis and Septic Shock: A Retrospective Before-After Study. Chest. 2017 Jun;151(6):1229-1238. doi: 10.1016/j.chest.2016.11.036. Epub 2016 Dec 6. PMID 27940189
- [Background] Marik PE. The physiology of volume resuscitation. Curr Anesthesiol Rep 2014; 4:353-59.
- [Background] Marik PE. Iatrogenic salt water drowning and the hazards of a high central venous pressure. Ann Intensive Care. 2014 Jun 21;4:21. doi: 10.1186/s13613-014-0021-0. eCollection 2014. PMID 25110606
- [Background] Marik P, Bellomo R. A rational approach to fluid therapy in sepsis. Br J Anaesth. 2016 Mar;116(3):339-49. doi: 10.1093/bja/aev349. Epub 2015 Oct 27. PMID 26507493
- [Background] Marik PE. Fluid Responsiveness and the Six Guiding Principles of Fluid Resuscitation. Crit Care Med. 2016 Oct;44(10):1920-2. doi: 10.1097/CCM.0000000000001483. No abstract available. PMID 26571187
- [Background] Monnet X, Marik PE, Teboul JL. Prediction of fluid responsiveness: an update. Ann Intensive Care. 2016 Dec;6(1):111. doi: 10.1186/s13613-016-0216-7. Epub 2016 Nov 17. PMID 27858374
- [Background] Marik PE, Linde-Zwirble WT, Bittner EA, Sahatjian J, Hansell D. Fluid administration in severe sepsis and septic shock, patterns and outcomes: an analysis of a large national database. Intensive Care Med. 2017 May;43(5):625-632. doi: 10.1007/s00134-016-4675-y. Epub 2017 Jan 27. PMID 28130687
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605
- [Background] ProCESS Investigators; Yealy DM, Kellum JA, Huang DT, Barnato AE, Weissfeld LA, Pike F, Terndrup T, Wang HE, Hou PC, LoVecchio F, Filbin MR, Shapiro NI, Angus DC. A randomized trial of protocol-based care for early septic shock. N Engl J Med. 2014 May 1;370(18):1683-93. doi: 10.1056/NEJMoa1401602. Epub 2014 Mar 18. PMID 24635773
- [Background] Mouncey PR, Osborn TM, Power GS, Harrison DA, Sadique MZ, Grieve RD, Jahan R, Harvey SE, Bell D, Bion JF, Coats TJ, Singer M, Young JD, Rowan KM; ProMISe Trial Investigators. Trial of early, goal-directed resuscitation for septic shock. N Engl J Med. 2015 Apr 2;372(14):1301-11. doi: 10.1056/NEJMoa1500896. Epub 2015 Mar 17. PMID 25776532
- [Background] ARISE Investigators; ANZICS Clinical Trials Group; Peake SL, Delaney A, Bailey M, Bellomo R, Cameron PA, Cooper DJ, Higgins AM, Holdgate A, Howe BD, Webb SA, Williams P. Goal-directed resuscitation for patients with early septic shock. N Engl J Med. 2014 Oct 16;371(16):1496-506. doi: 10.1056/NEJMoa1404380. Epub 2014 Oct 1. PMID 25272316
- [Background] de Azevedo JR, Torres OJ, Beraldi RA, Ribas CA, Malafaia O. Prognostic evaluation of severe sepsis and septic shock: procalcitonin clearance vs Delta Sequential Organ Failure Assessment. J Crit Care. 2015 Feb;30(1):219.e9-12. doi: 10.1016/j.jcrc.2014.08.018. Epub 2014 Sep 10. PMID 25241933
- [Background] Ruiz-Rodriguez JC, Caballero J, Ruiz-Sanmartin A, Ribas VJ, Perez M, Boveda JL, Rello J. Usefulness of procalcitonin clearance as a prognostic biomarker in septic shock. A prospective pilot study. Med Intensiva. 2012 Oct;36(7):475-80. doi: 10.1016/j.medin.2011.11.024. Epub 2012 Jan 16. PMID 22257436
- [Background] Flannery AH, Adkins DA, Cook AM. Unpeeling the Evidence for the Banana Bag: Evidence-Based Recommendations for the Management of Alcohol-Associated Vitamin and Electrolyte Deficiencies in the ICU. Crit Care Med. 2016 Aug;44(8):1545-52. doi: 10.1097/CCM.0000000000001659. PMID 27002274
- [Background] Mancl EE, Muzevich KM. Tolerability and safety of enteral nutrition in critically ill patients receiving intravenous vasopressor therapy. JPEN J Parenter Enteral Nutr. 2013 Sep;37(5):641-51. doi: 10.1177/0148607112470460. Epub 2012 Dec 27. PMID 23270986
- [Background] Russell JA, Walley KR, Singer J, Gordon AC, Hebert PC, Cooper DJ, Holmes CL, Mehta S, Granton JT, Storms MM, Cook DJ, Presneill JJ, Ayers D; VASST Investigators. Vasopressin versus norepinephrine infusion in patients with septic shock. N Engl J Med. 2008 Feb 28;358(9):877-87. doi: 10.1056/NEJMoa067373. PMID 18305265
- [Background] Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med. 1985 Oct;13(10):818-29. PMID 3928249
- [Background] Zimmerman JE, Kramer AA, McNair DS, Malila FM. Acute Physiology and Chronic Health Evaluation (APACHE) IV: hospital mortality assessment for today's critically ill patients. Crit Care Med. 2006 May;34(5):1297-310. doi: 10.1097/01.CCM.0000215112.84523.F0. PMID 16540951
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Background] Ferreira FL, Bota DP, Bross A, Melot C, Vincent JL. Serial evaluation of the SOFA score to predict outcome in critically ill patients. JAMA. 2001 Oct 10;286(14):1754-8. doi: 10.1001/jama.286.14.1754. PMID 11594901
- [Derived] Iglesias J, Vassallo AV, Patel VV, Sullivan JB, Cavanaugh J, Elbaga Y. Outcomes of Metabolic Resuscitation Using Ascorbic Acid, Thiamine, and Glucocorticoids in the Early Treatment of Sepsis: The ORANGES Trial. Chest. 2020 Jul;158(1):164-173. doi: 10.1016/j.chest.2020.02.049. Epub 2020 Mar 17. PMID 32194058

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between February 14th, 2018 and April 29th, 2019, 256 patients were evaluated within two community hospital intensive care units.
Pre-assignment Details: Patients excluded from enrollment based on their diagnosis upon admission (ineligible unless they were admitted to the ICU for sepsis, 33 patients), end stage disease (20), had a DNR/DNI (17), or required immediate surgery (11).
Period: Overall Study
Arm/Group | Treatment Arm | Placebo Arm
Started | 70 | 70
Completed | 68 | 69
Not Completed | 2 | 1
Not completed — Exclusion due to terminal disease | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment: Based on published clinical data, vitamin C pharmacokinetic modeling, the package insert as well as the preliminary study by Marik et al, Vitamin C will be administered as an intravenous dose of 6gm per day divided in 4 equal doses. This dosage is reported to be devoid of any complications or side effects. Hydrocortisone will be dosed according to the consensus guidelines of the American College of Critical Care Medicine. Thiamine will be administered according to current recommendations in a dose of 200mg q 12 hourly. This will be continued for 4 days, or less if discharged from the ICU prior.
  Ascorbic Acid: Ascorbic Acid 1.5g IV piggyback every 6 hours for 4 days (or discharge from ICU if prior to 4 days).
  Thiamine: Thiamine 200mg IV piggyback every 12 hours for 4 days (or discharge from ICU if prior to 4 days).
  Hydrocortisone: Hydrocortisone 50mg IV push every 6 hours for 4 days (or discharge from ICU if prior to 4 days).
- Comparator: Vitamin C placebo will consist of an identical bag of 100mL normal saline (but with no vitamin C) and will be labeled "Vitamin C or Placebo". Placebo will be infused over 30 minutes as per the infusion instructions of the active vitamin and protected from light with a brown bag. Hydrocortisone placebo will be provided as an identical 3mL syringe as 1mL of normal saline.The thiamine placebo will be placed in a 50mL bag of Normal Saline labeled "Thiamine 200mg or Placebo" and run over 30 minutes (100mL/hr) Placebo patients will receive a matching 50mL bag of Normal Saline. All of these will be given for up to 4 days, or less if discharged from the ICU prior.
  Sodium Chloride 0.9%: Placebo "Ascorbic Acid" 100mL IV piggyback every 6 hours, Placebo "Thiamine" 50mL IV piggyback every 12 hours, and Placebo "Hydrocortisone" IV push every 6 hours for 4 days (or discharge from ICU if prior to 4 days).
- Total: Total of all reporting groups
Arm/Group | Treatment | Comparator | Total
Number analyzed (Participants) | 68 | 69 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (12) | 67 (14) | 68 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 42 | 78
  Male | 32 | 27 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 66 | 65 | 131
  Non-Caucasian | 2 | 4 | 6
Comorbidities [Count of Participants; unit: Participants]
  Coronary Artery Disease (CAD) | 25 | 21 | 46
  Diabetes | 24 | 33 | 57
  Dementia | 7 | 4 | 11
  Heart failure | 18 | 13 | 31
  Malignancy | 15 | 11 | 26
  Chronic Obstructive Pulmonary Disease (COPD) | 23 | 17 | 40
  Cirrhosis | 0 | 3 | 3
  End Stage Renal Disease (ESRD) | 3 | 0 | 3
  Chronic Kidney Disease (CKD) | 10 | 4 | 14
  Morbid Obesity (BMI >40) | 16 | 13 | 29
  Immunocompromised | 6 | 5 | 11
Primary diagnosis [Count of Participants; unit: Participants]
  Pneumonia | 29 | 30 | 59
  Urinary tract infection | 18 | 25 | 43
  Primary bacteremia | 9 | 11 | 20
  Gastrointestinal/biliary | 9 | 8 | 17
  Other | 13 | 9 | 22
Other Baseline Characteristics [Count of Participants; unit: Participants]
  Need for mechanical ventilation | 34 | 35 | 69
  Vasopressor usage during hospital admission | 56 | 47 | 103
  Acute Kidney Injury (Stage 1 or higher based on KDIGO definitions) | 54 | 52 | 106
  Positive blood cultures | 22 | 23 | 45
Baseline Labs [Mean (Standard Deviation); unit: mg/dL]
  Creatinine (mg/dL) | 2.1 (1.5) | 2 (1.51) | 2 (0)
  Ascorbic acid level (mg/dL) | 0.52 (1) | 0.48 (0.4) | 0.5 (0)
  Thiamine (mg/dL) | 193 (144) | 148 (53) | 170 (0)
Baseline White Blood Cell Count (WBC) x10^9/L [Mean (Standard Deviation); unit: x10^9 cells/L] | 16 (10) | 19 (9.7) | 17.5 (0)
Baseline Lactate (mM/L) [Mean (Standard Deviation); unit: mM/L] | 4.45 (3.5) | 4.8 (4.2) | 4.6 (0)
Baseline Procalcitonin (ng/mL) [Mean (Standard Deviation); unit: ng/mL] | 44 (72) | 23 (38) | 33.5 (0)
Baseline Sequential Organ Failure Assessment (SOFA) Score [Mean (Standard Deviation); unit: scores on a scale] — Score from 0 to 24, with 24 indicating more organ dysfunction
  scores on a scale | 8.3 (3) | 7.9 (3.5) | 8.1 (0)
Acute Physiology And Chronic Health Evaluation (APACHE) II [Mean (Standard Deviation); unit: scores on a scale] — Score from 0 to 71, with a higher score indicating increased risk of ICU mortality
  scores on a scale | 24 (7.6) | 24.9 (8.7) | 24.5 (0)
Acute Physiology And Chronic Health Evaluation (APACHE) IV [Mean (Standard Deviation); unit: scores on a scale] — Score from 0 to 93, with a higher score indicating increased risk of ICU mortality
  scores on a scale | 88 (28.3) | 87.5 (29.7) | 87.8 (0)
APACHE IV predicted mortality (%) [Mean (Standard Deviation); unit: percentage of predicted mortality] — Percentage of predicted mortality as derived from APACHE IV score
  percentage of predicted mortality | 34 (3) | 33.6 (2.6) | 33.8 (0)

OUTCOME MEASURES:

1. Primary Outcome: Time to Vasopressor Independence (Hours)
Description: Defined as the time from starting the active treatment/placebo to discontinuation of all pressors.
Time Frame: From start of vasopressor medication to final discontinuation of vasopressor medication, up to 7 days.
Population: Patients on vasopressor therapy in each group.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- HAT Treatment: Receiving Hydrocortisone, Ascorbic Acid, and Thiamine
- Comparator: Receiving placebo
Arm/Group | HAT Treatment | Comparator
Number analyzed (Participants) | 60 | 57
hours | 27 (22) | 53 (38)
Statistical Analysis 1: Comparison: HAT Treatment vs Comparator; Test type: Non-Inferiority — Based on the results of the preliminary study of Marik et al, 5 we projected that the combination of ascorbic acid, thiamine, and hydrocortisone could reduce time to vasopressor discontinuation from 54 (+/-30 hours) vs 30 hours. For the additional primary outcome, we projected a greater change of SOFA score of 4 (+/-3) vs 2. Assuming a type 1 error of 5% (alpha of 0.05) and a power of 80%, this study would require a sample size of 94 patients; p < 0.001, t-test, 2 sided

2. Primary Outcome: Change in Sequential Organ Failure Assessment (SOFA) Score
Description: Defined as the day 4 post-randomization SOFA score minus the initial SOFA score. The Sequential Organ Failure Assessment (SOFA) Score is a mortality prediction score that is based on the degree of dysfunction of six organ systems. The score is calculated on admission and every 24 hours until discharge using the worst parameters measured during the prior 24 hours SOFA score ranges from 0 (no organ dysfunction) to 24 (highest possible score / organ dysfunction).
Time Frame: 4 days post-randomization
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 68 | 69
score on a scale | 2.9 (3.3) | 1.93 (3.5)

3. Secondary Outcome: Procalcitonin (PCT) Clearance
Description: PCT at 96 hours minus initial PCT, divided by the initial PCT multiplied by 100.
Time Frame: 4 days post-randomization
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 68 | 69
Percent | 63 (170) | 58 (66)

4. Secondary Outcome: ICU Mortality
Description: ICU mortality rate
Time Frame: From admission to hospital until final discharge from the ICU, up to 28 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 68 | 69
Participants | 6 | 10

5. Secondary Outcome: ICU Length of Stay
Description: Time from admitting to ICU to discharge.
Time Frame: From admission to the ICU until final discharge from the ICU, up to an average of 7 days.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 68 | 69
days | 4.76 (4.3) | 4.66 (3.45)

6. Secondary Outcome: Ventilator Free Days
Description: Number of days alive and off of the ventilator at day 28.
Time Frame: 28 Days post-randomization
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 68 | 69
Days | 22 (6.2) | 22.4 (4.3)

7. Secondary Outcome: Hospital Length of Stay
Description: Time from admitting to discharge of hospital stay.
Time Frame: From admission to the hospital until final discharge, up to 28 days.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 68 | 69
Days | 11.5 (6.8) | 11 (6.2)

8. Secondary Outcome: Hospital Mortality
Description: In-hospital mortality rate.
Time Frame: Survival until hospital discharge, up to 28 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Placebo Arm
Number analyzed (Participants) | 68 | 69
Participants | 11 | 13

ADVERSE EVENTS:
Time Frame: Each participant was assessed for adverse events up to hospital discharge, or up to 28 days.
Arm/Group | Treatment Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 11/68 | 13/69
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/69
Other Adverse Events (participants affected / at risk) | 0/68 | 0/69

LIMITATIONS AND CAVEATS:
The relative weakness was its small, homogenous (primarily caucasian) cohort size, limiting the ability to detect differences in hospital mortality and length of stay.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/59/NCT03422159/Prot_003.pdf
  • Statistical Analysis Plan (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/59/NCT03422159/SAP_006.pdf
  • Informed Consent Form (2018-05-31): https://cdn.clinicaltrials.gov/large-docs/59/NCT03422159/ICF_005.pdf